CLINICAL TRIAL: NCT07328126
Title: Effect of Muscle Energy Technique on Latissimus Dorsi on Pain , Functional Disability and Range of Motion in Patients With Mechanical Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/07
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-10

CONDITIONS: Mechanical Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative physical therapy (Active Comparator): Hot pack + TENS (10 min), followed by a structured program of warm-up, 20-minute core/back strengthening, stretching (hip flexors, hamstrings, lumbar extensors), and cool-down exercises.
  Interventions: Procedure: Conservative physical therapy
- Post facilitation stretch of latissimus dorsi with conservative physical therapy (Experimental): Receives the same conservative physical therapy as the control group plus Latissimus Dorsi Muscle Energy Technique (isometric contraction for 10seconds, relaxation 2-3seconds, followed by 10seconds stretch, applied bilaterally each session).
  Interventions: Procedure: Post-facilitation stretch of latissimus dorsi with conservative physical therapy

INTERVENTIONS:
Procedure: Conservative physical therapy — Hot pack + TENS (10 min), followed by a structured program of warm-up, 20-minute core/back strengthening, stretching (hip flexors, hamstrings, lumbar extensors), and cool-down exercises.
  Arms: Conservative physical therapy
Procedure: Post-facilitation stretch of latissimus dorsi with conservative physical therapy — Receives the same conservative physical therapy as the control group plus Latissimus Dorsi Muscle Energy Technique (isometric contraction for 10seconds, relaxation 2-3seconds, followed by 10seconds stretch, applied bilaterally each session).
  Arms: Post facilitation stretch of latissimus dorsi with conservative physical therapy

SUMMARY:
Mechanical low back pain (LBP) stems from spinal structures or surrounding tissues, often caused by overuse or trauma, and is prevalent globally with high recurrence rates. Key contributing factors include biomechanical, psychological, and social elements. The latissimus dorsi (LD), along with other back muscles, plays a crucial role in lumbar stability via the thoracolumbar fascia. Stretching the LD has shown positive effects in reducing pain and improving function in chronic LBP patients. Physical therapy treatments include manual therapy, core stabilization, and flexibility exercises. Muscle Energy Techniques (MET), particularly targeting the LD, can enhance flexibility and spinal mobility when applied correctly.

DETAILED DESCRIPTION:
Mechanical low back pain (MLBP) originates from structural components of the spine, such as intervertebral discs, muscles, ligaments, or joints, and is commonly caused by repetitive trauma, poor posture, or overuse. It is a leading cause of functional disability worldwide, with high recurrence rates. Physiotherapy plays a central role in managing MLBP by addressing contributing biological, psychological, and social factors. The latissimus dorsi (LD) muscle, due to its anatomical connection with the pelvis via the thoracolumbar fascia (TLF), significantly influences lumbar stability. Impaired extensibility or overactivity of the LD can contribute to mechanical dysfunction. Incorporating LD stretching into rehabilitation protocols has shown enhanced outcomes in pain reduction and functional improvement. Muscle Energy Techniques (MET), particularly Post Facilitation Stretching, utilize controlled muscle contractions to improve flexibility and relieve tension in shortened muscles. Proper application of MET targeting the LD has demonstrated effectiveness in increasing range of motion and supporting spinal stability in patients with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients had low back pain for more than 3 months Moderate disability (20 to 40 %) determined through Oswestry Disability Index Subjects with pain ranging 3 to 8 on NPRS Able to perform ROM of lumbar spine (flexion and extension) within range of pain Patient were not under any medical treatment (analgesics etc) both male and female

Exclusion Criteria:

* presence of any red flags (i.e tumor , metabolic disease, rheumatoid arthritis , osteoporosis , history of use of steroids ) SLR test positive Muscle weakness or paralysis of lower extremity Prior surgery of lumbar spine and pregnancy Any psychological problem

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Low back pain | 4 weeks
  Numeric Pain Rating Scale will be used. An 11-point scale comprising a number from 0 through 10; 0 indicates "no pain", and 10 indicates the "worst imaginable pain". Patients are instructed to choose a single number from the scale that best indicates their level of pain.
Functional Disability of back | 4 weeks
  Oswestry disability index will be used. To evaluate the functional impact of low back pain on a person's daily life.
  It consists of 10 items on the degree of severity to which back (or leg) trouble has affected the ability to manage in everyday life. The 10 sections cover the pain and the daily function (including pain intensity, personal hygiene, lifting, walking, sitting, standing, sleeping, sexual activity, social activity, and traveling). Each item is rated on a 6-point scale (0-5); the higher score means the higher level of disability related to LBP. The present study used the traditional Chinese version of the ODI 2.1
Range of motion of low back. | 4 weeks
  Dual Inclinometer will be used. It is a handheld, circular, fluid-filled disc that has a weighted gravity pendulum attached to it that is maintained in the vertical direction. It is graduated by 0.5 degree intervals over 360.

CONTACTS AND LOCATIONS:
Overall Officials: Laraib Khurshid, DPT, Principal Investigator — Foundation University Islamabad
Locations (1):
- Foundation University Islamabad, Rawalpindi, Punjab Province, Pakistan